CLINICAL TRIAL: NCT03243526
Title: The Effect of Fluid Management Guided by Pulse Pressure Variation Versus Central Venous Pressure on Extra Vascular Lung Water Assessed by Lung Ultrasound Score During Liver Transplantation. A Randomized Controlled Trial.
Brief Title: Effect of Fluid Management Guided by Pulse Pressure Variation Vs Central Venous Pressure on Lung Water Assessed by Lung Ultrasound During Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Elayashy Mohamed Ahmed Hassan, clinical professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-42-2017
Record Dates: First submitted 2017-07-27; First posted 2017-08-09 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Lung; Congestive; Liver Transplantation
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: two groups one recieve fluid guided by CVP and othe by PPV
Who Masked: Participant, Outcomes Assessor
Masking Description: patient will be blinded and person who will do lung ultrasound
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Central venous pressure group (Placebo Comparator): fluid therapy to maintain CVP not 5 cmH2o
  Interventions: Other: fluid therapy
- Pulse pressure variation (Experimental): fluid therapy will be guided by PPV to be less than 14%
  Interventions: Other: fluid therapy

INTERVENTIONS:
Other: fluid therapy — fluid resuscitation guided by CVP or PPV

SUMMARY:
the aim in this study to assess the effect of fluid management in patient undergoing orthotopic liver transplantation either by using pulse pressure variation or by central venous pressure. we will assess the impact of fluid management by either methods on oxygenation and extra vascular lung water visualized by lung ultrasound.

DETAILED DESCRIPTION:
After induction of anesthesia lung ultrasound will be performed and arterial blood gases (ABG) will be taken.

All patients in both groups will receive maintenance fluid in the form of crystalloids (ringer acetate) 4 ml/kg/H. Then fluid boluses will be given according to each group:

Group c (cvp): will receive 250 ml albumin 5% boluses to maintain CVP around 5 cmH2o Group P (ppv): will receive 250 ml albumin 5% boluses to maintain PPV below 13% as detected from invasive blood pressure monitor.

For all patients in both groups: blood transfusion will be indicated with decreased HB% level below 7 mg/dl in arterial blood gases. Other blood product (FFP, platelets and cryoprecipitate) transfusion will be guided by lab results and clinical status of patient. Plasma will be transfused if INR > 1.5 and platelets will be transfused if count < 50, 000

Lung ultrasound will be performed to diagnose EVLW. A Philips C5 ultrasound system (frequency 5Hz; Philips Medical Systems, Suresnes, France) with an ordinary echo probe will be used. Chest ultrasound will be performed using the 12 regions method. Intercostals spaces on each side will be examined anteriorly (midclavicular line), laterally (anterior axillary line) and posteriorly (posterior axillary line) Four ultrasound aeration patterns a. Normal aeration (N): 0 score ; line sliding sign associated with respiratory movement or less than 3 B lines ; b. Moderate loss of lung aeration: score 1 ; a clear number of multiple visible B-lines with horizontal spacing between adjacent B lines ≤ 7 mm (B7 lines) c. Severe loss of lung aeration: score 2; multiple B lines fused together that were difficult to count with horizontal spacing between adjacent B lines ≤ 3 mm (B3 lines); and d. Pulmonary consolidation: score 3; hyperechoic lung tissue, accompanied by dynamic air bronchogram.

The final LUS of the patient was the sum of each regional ultrasound score (ranging from 0 to 36).

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status II- IV
2. Child C (end stage liver disease) ESLD patient.
3. Age (18- 70) years
4. Patients undergoing orthotopic liver transplantation.

Exclusion Criteria:

1. Parents' refusal.
2. Patients with chronic pulmonary disease ( Asthma, obstructive lung disease or restrictive lung diseases)
3. Patient with impaired diastolic function more than grade I.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
lung ultrasound score | 5 minutes after surgical wound closure
  lung score assessed by lung ultrasound to assess lung water. score range from 0 to 36

SECONDARY OUTCOMES:
lung ultrasound score | baseline 10 minutes after induction. and 1 hour after Intensive care admission
  lung score assessed by lung ultrasound to assess lung water. score range from 0 to 36
P/F ratio | baseline 10 min after induction, 5 minutes after surgical wound closure and 1 hour after intensive care admission
  ratio of Po2 to fraction of inspired oxygen.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital , Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fallon MB, Abrams GA. Pulmonary dysfunction in chronic liver disease. Hepatology. 2000 Oct;32(4 Pt 1):859-65. doi: 10.1053/jhep.2000.7519. No abstract available. PMID 11003635
- [Background] Bozbas SS, Eyuboglu FO, Ozturk Ergur F, Gullu Arslan N, Sevmis S, Karakayali H, Haberal M. Pulmonary complications and mortality after liver transplant. Exp Clin Transplant. 2008 Dec;6(4):264-70. PMID 19338487
- [Background] Gardelli G, Feletti F, Nanni A, Mughetti M, Piraccini A, Zompatori M. Chest ultrasonography in the ICU. Respir Care. 2012 May;57(5):773-81. doi: 10.4187/respcare.01743. PMID 22546298
- [Background] Aghdashi M, Broofeh B, Mohammadi A. Diagnostic performances of high resolution trans-thoracic lung ultrasonography in pulmonary alveoli-interstitial involvement of rheumatoid lung disease. Int J Clin Exp Med. 2013 Aug 1;6(7):562-6. Print 2013. PMID 23936595